CLINICAL TRIAL: NCT00378183
Title: A Randomized Open-Label, Rater Blinded Assessment of Optimal Treatment Change Strategy to Risperidone for Patients Intolerant of Olanzapine
Brief Title: A Study Comparing Three Strategies to Switch Patients With Schizophrenia or Schizoaffective Disorder to Risperidone After Unsuccessful Treatment With Olanzapine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012520
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: weight loss; behavioral therapy; risperidone; switching antipsychotics; schizoaffective disorder; Risperdal; schizophrenia; olanzapine; Zyprexa
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Weight Loss | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to compare three strategies for switching patients with schizophrenia or schizoaffective disorder to the atypical antipsychotic, risperdone, after they have been unsuccessfully treated with another atypical antipsychotic, olanzapine. In the second phase of this study, investigators will assess the effectiveness of behavioral therapy in reducing body weight in risperdone-treated patients who are overweight or have problems with diabetes or blood sugar.

DETAILED DESCRIPTION:
Data regarding the safety and effectiveness of different strategies for switching subjects with schizophrenia from one antipsychotic medication to another are very rare. Studies that have examined various switching designs, especially with regard to the newer atypical antipsychotic agents, suggest that either abrupt or gradual discontinuation does not inevitably lead to worsening of symptoms. This study is randomized (patients are assigned different treatments based on chance), open-label, with a parallel group design to assess the safety and effectiveness of each of three strategies of discontinuing olanzapine and starting risperidone. The first strategy is the discontinuation of olanzapine on the day risperidone is started. The second strategy involves a reduction in the dose of olanzapine to one half of the study entry dose on the day risperidone is started. The reduced dose of olanzapine is to be given for one week and then discontinued. In the third strategy, the dose of olanzapine remains unchanged for the first week, then is reduced by one half of the study entry dose, and at the end of the second week is discontinued. In all three strategies, patients take the same dose of risperidone: 1 mg by mouth twice a day for 3 days, then 2 mg twice a day for the next 4 days. Further increase or decrease of risperidone dose and/or changing to a single daily dose can be carried out at the end of the first week. Additionally, after 6 weeks of risperidone therapy, patients who are overweight or have problems with diabetes or blood sugar may enter a second phase of the study that examines weight loss. In this phase, patients are randomized to receive routine clinical care or training on weight management behavioral techniques while continuing to take risperidone for an additional 14 weeks. At the end of 14 weeks, total weight loss, changes in lipids, cholesterol and other laboratory measures will be compared between the two groups. The study hypothesis is that symptom improvement or worsening at week 14, as measured by total score on the Positive and Negative Syndrome Scale (PANSS), should not differ depending on the method of switching from olanzapine to risperidone. Safety evaluations incude collection of adverse events, clinical laboratory tests and assessment of vital signs.

The patients will receive oral tablets of risperidone 1 to 2 milligram[mg] twice a day (higher or lower dose and/or changing to single daily dose allowed at end of the first week) for the duration of 6 weeks in phase 1, and then for 14 more weeks in phase 2 of the study. Olanzapine: none; or half of the study entry dose for 1 week; or study entry dose for 1 week, then half of the study entry dose for an additional week.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) diagnosis of schizophrenia or schizoaffective disorder
* Taking a stable dose of olanzapine for at least 30 days
* Have not experienced an acute exacerbation of their psychotic symptoms in the preceding 3 months
* Either had only a marginal clinical response to olanzapine, or had unacceptable side effects related to weight gain including obesity, diabetes or abnormal glucose metabolism

Exclusion Criteria:

* Patients with a history of treatment failure with, or significant adverse events attributable to, risperidone, or known sensitivity to risperidone
* A history of antipsychotic therapy other than olanzapine in the 30 days preceding randomization
* Presence of serious or unstable illnesses: liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, psychiatric or metabolic disturbances
* Diagnosis of substance dependence
* Pregnant or nursing female, or those lacking adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-02; Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
The change in total Positive and Negative Syndrome Scale (PANSS) score from baseline at week 14 of Phase 2.

SECONDARY OUTCOMES:
The change from baseline in Client Satisfaction Questionnaire (CSQ-8) score at week 14 of Phase 2 and the change from baseline in Global Assessment of Functioning (GAF) score at week 14 of Phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Derived] Ganguli R, Brar JS, Mahmoud R, Berry SA, Pandina GJ. Assessment of strategies for switching patients from olanzapine to risperidone: a randomized, open-label, rater-blinded study. BMC Med. 2008 Jun 30;6:17. doi: 10.1186/1741-7015-6-17. PMID 18590519